CLINICAL TRIAL: NCT05064046
Title: Educating Providers About Health Disparities in Lung Cancer Screening
Brief Title: Educating Providers About Lung Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00003967; 3R01CA207228-05S1 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
Keywords: lung cancer screening; provider education; health disparities
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Arm 1- LuCa + Health Disparity module: Providers enrolled in the LuCa+ arm will complete lesson 1 of the LuCa training and complete the Health Disparity module. Arm 2- LuCa module: Providers enrolled in the LuCa arm will complete session 1 of the LuCa training.
Who Masked: Investigator
Masking Description: The research investigators will be blinded from the study arm of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LuCa + Health Disparity module (Experimental): Participants will be asked to complete the Health Disparities module that is an interactive CME/CE online course which offers 0.5 continuing education credit hours.
  The will also be asked to complete the LuCa course.
  Interventions: Behavioral: LuCa + Health Disparity module
- LuCa only module (Active Comparator): LuCa is a free interactive CME/CE online course entitled, "Lung Cancer and the Primary Care Provider". For the purpose of this study, participants will be asked to complete session 1 which offers 1.0 continuing education credit hours, including AMA PRA Category 1 credits, AANP, and AAFP Prescribed credits.
  Interventions: Behavioral: LuCa + Health Disparity module

INTERVENTIONS:
Behavioral: LuCa + Health Disparity module — The Health Disparity course will review disparities in the burden of lung cancer across racial/ethnic groups, discuss differences in smoking patterns and use of evidence-based smoking cessation, and describe emerging disparities in lung cancer screening. The course will also offer resources for providers to address common barriers to screening among underserved/underrepresented groups, including insurance information, transportation options, procedure time, and patient navigation assistance.
  Lesson 1 of the LuCa online course addresses lung cancer screening and shared decision making.

SUMMARY:
We are conducting a randomized trial to compare the Health Disparities module to an existing provider module on lung cancer screening to evaluate the impact on primary care providers' knowledge, attitudes, and lung cancer screening referrals of African American and White patients.

DETAILED DESCRIPTION:
We are conducting a randomized trial of two online, provider-facing education modules regarding lung cancer screening and smoking cessation. We will accrue 70 MedStar primary care providers (PCP). The baseline survey will incorporate items regarding lung cancer screening knowledge, providers' attitudes towards lung cancer screening, lung cancer screening ordering practices and provider characteristics. At the end of the baseline survey, PCPs will be randomly assigned to the LuCa + Health Disparities or LuCa only. PCPs will be asked to complete the intervention and the post-test within 1 week of randomization. The post test will cover knowledge of lung cancer screening, attitudes and opinions toward LCS. To assess PCP lung cancer screening ordering practices, we will review the MedConnect Electronic Health Record (EHR) to compare the two study groups post-randomization on the number of orders made for LCS.

ELIGIBILITY:
Inclusion Criteria:

* MedStar provider (attending or resident physician, physician's assistant, or nurse practitioner)
* English speaking
* ability to provide meaningful consent
* ability to provide last two digits of NPI.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Number of providers with improved mean lung cancer screening knowledge score | 1 week
  Knowledge about lung cancer screening
Number of providers with improved mean attitudes score | 1 week
  Attitudes about lung cancer screening

SECONDARY OUTCOMES:
Rate of lung cancer screening referrals | 2 months post-randomization
  Lung cancer screening referrals from the electronic health record

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Health Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith L, Williams RM, Whealan J, Windels A, Anderson ED, Parikh V, Breece CJ, Puran N, Shepherd AK, Geronimo M, Luta G, Adams-Campbell L, Taylor KL. Development and Evaluation of Brief Web-Based Education for Primary Care Providers to Address Inequities in Lung Cancer Screening and Smoking Cessation Treatment. J Cancer Educ. 2023 Aug;38(4):1296-1303. doi: 10.1007/s13187-023-02262-3. Epub 2023 Jan 13. PMID 36637713